CLINICAL TRIAL: NCT05654259
Title: Obesity and Sleep Apnea in Pregnancy
Brief Title: Obesity and OSA in Pregnancy
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Qi Fu, Professor-Internal Medicine, University of Texas Southwestern Medical Center
Other Study IDs: STU 062018-089
Record Dates: First submitted 2022-12-08; First posted 2022-12-16 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Obesity; Obesity, Maternal; Obstructive Sleep Apnea; Blood Pressure
Keywords: obesity; pregnancy; sleep apnea; blood pressure
MeSH Terms: conditions — Obesity; Pregnancy in Obesity; Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- obese women with normal gestational weight gain: obese women (body mass index ≥30 kg/m2) with weight gain 5-9 kg
- obese women excessive gestational weight gain: obese women (body mass index ≥30 kg/m2) with weight gain >9 kg
- non-obese women with normal gestational weight gain: non-obese women (body mass index 18.5-24.9 kg/m2) with weight gain 11.5-16 kg
- non-obese women with excessive weight gain: non-obese women (body mass index 18.5-24.9 kg/m2) with weight gain >16 kg
- obese women with OSA: obese women (body mass index ≥30 kg/m2) with Obstructive Sleep Apnea (OSA) (Apnea and Hypopnea Index (AHI) ≥5 events/hr
- obese women without OSA: obese women (body mass index ≥30 kg/m2) without Obstructive Sleep Apnea (OSA) (AHI <5 events/ hr)
- non-obese women without OSA: non-obese women without OSA (AHI <5 events/ hr)

SUMMARY:
The purposes of this project are 1) to compare the impact of maternal obesity versus excessive gestational weight gain on obstructive sleep apnea (OSA) in obese and non-obese women; 2) to investigate the mechanism(s) by which obesity and OSA increase cardiovascular risk during pregnancy; and 3) to identify biomarker(s) for obesity-related OSA in pregnant women.

DETAILED DESCRIPTION:
Aim 1: To test the hypothesis that maternal obesity increases OSA risk but to a greater extent in obese women with excessive gestational weight gain vs. obese women with normal weight gain vs. non-obese women with excessive weight gain. Study team will enroll early pregnant (≤12 weeks of gestation) obese (pre-pregnancy body mass index ≥30 kg/m2) and non-obese (body mass index 18.5-24.9 kg/m2) women and follow participants throughout gestation. In-home sleep testing will be carried out during all phases of pregnancy: early pregnancy (4-12 weeks gestation), late pregnancy (30-34 weeks of gestation) and postpartum (6-10 weeks after delivery). Investigator will compare AHI (primary endpoint), the development or worsening of OSA, and pregnancy outcomes in obese and non-obese women with and without weight gain above the Institute of Medicine (IOM) recommended levels. Various body composition areas, (e.g., neck, waist, or hips) that may be associated with risk for sleep apnea will also be measured.

Aim 2: To test the hypothesis that obesity is associated with sympathetic activation, while OSA magnifies this abnormality during pregnancy. Study team will use the state-of-the-art technique of microneurography to measure resting sympathetic activity (primary endpoint) and sympathetic neural responses to physiological stimulations (e.g., mental stress, exercise and upright posture) during early (<12 weeks) and late (30-34 weeks) pregnancy, and postpartum (6-10 weeks post) in obese women with and without OSA and non-obese women without OSA.

Aim 3: To test the hypothesis that corin content is greater in obese than nonobese women during pregnancy, and it is the greatest in obese pregnant women with OSA. Venous blood samples will be taken in women enrolled in Aim 2 study for measurements of serum corin content (primary endpoint) and pregnancy-specific angiogenic factors such as soluble fms-like tyrosine kinase 1, placental growth factor, and soluble endoglin. The relationships between maternal corin content, pregnancy-specific angiogenic factors, sympathetic activity, and BP will be explored.

ELIGIBILITY:
Inclusion Criteria:

* Both obese and non-obese (normal weight) early pregnant women aged ≥18 years old will be permitted to participate in this project.
* No restriction with respect to race and socioeconomic status
* Women with a prior history of complicated pregnancy (i.e., gestational hypertension, preeclampsia, HELLP syndrome, gestational diabetes, preterm birth, intrauterine growth restriction, etc.) will be allowed to participate.
* Obese women with previously diagnosed OSA will be allowed to participate if they are not currently on any recognized treatments such as Continuous Positive Airway Pressure (CPAP), oral appliances or nasal expiratory positive airway pressure.
* Those who have had surgery for OSA in the past will be excluded.
* Women taking low-dose aspirin will be allowed to participate in this project.

Exclusion Criteria:

* Current multiple pregnancy;
* Known major fetal chromosomal or anatomical abnormalities;
* Recurrent miscarriage (three or more);
* Chronic essential hypertension (systolic BP >140 mmHg and/or diastolic BP >90 mmHg);
* Any evidence of cardiovascular and pulmonary diseases by history or by physical examination;
* Kidney disease (serum creatinine >1.5 mg/dL);
* Coagulation disorders;
* Diabetes mellitus (fasting glucose ≥126 mg/dL or 2-hour oral glucose tolerance test glucose level ≥200 mg/dL) or other systemic illness;
* Any evidence of neurological disease;
* Psychiatric disease or psychological disorders;
* History of drug or alcohol abuse within the last 2 years; and
* Given the effects of exercise training on sympathetic neural control, endurance-trained athletes will be excluded. As this project focuses on sleep apnea in pregnancy, Women with other significant sleep disorders such as restless legs syndrome by Rest Leg Syndrome Diagnostic Index and insomnia by the Insomnia Severity Index or Pittsburgh Sleep Quality Index will be excluded; In addition, women who report taking a sleeping aid >1 time per month will be excluded.

Ages: 18 Years to 64 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — Study includes all women
Study Population: Obese and non-obese pregnant women with and without excessive gestational weight gain; Obese and non-obese pregnant women with and without OSA
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2018-07-11 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Apnea Hypopnea Index (AHI) | Early pregnancy (4-12 weeks gestation)
  The Apnea-Hypopnea Index or Apnoea-Hypopnoea Index (AHI) is an index used to indicate the severity of sleep apnea as measured by the Watch Pat device. It is represented by the number of apnea and hypopnea events per hour of sleep. The apneas (pauses in breathing) must last for at least 10 seconds and be associated with a decrease in blood oxygenation. A higher AHI value ≥5 indicates more severe sleep apnea
Apnea Hypopnea Index (AHI) | Late pregnancy (30-34 weeks of gestation)
  The Apnea-Hypopnea Index or Apnoea-Hypopnoea Index (AHI) is an index used to indicate the severity of sleep apnea as measured by the Watch Pat device. It is represented by the number of apnea and hypopnea events per hour of sleep. The apneas (pauses in breathing) must last for at least 10 seconds and be associated with a decrease in blood oxygenation. A higher AHI value ≥5 indicates more severe sleep apnea
Apnea Hypopnea Index (AHI) | Post partum (6-10 weeks after delivery)
  The Apnea-Hypopnea Index or Apnoea-Hypopnoea Index (AHI) is an index used to indicate the severity of sleep apnea as measured by the Watch Pat device. It is represented by the number of apnea and hypopnea events per hour of sleep. The apneas (pauses in breathing) must last for at least 10 seconds and be associated with a decrease in blood oxygenation. A higher AHI value ≥5 indicates more severe sleep apnea
Resting sympathetic activity | Early pregnancy (< 12 weeks gestation)
  Resting sympathetic activity is measured by microneurography, as expressed as the number of bursts per minute and as the number of bursts per 100 heart beats, to correct for differences in heart rate.
Resting sympathetic activity | Late pregnancy (30-34 weeks of gestation)
  Resting sympathetic activity is measured by microneurography, as expressed as the number of bursts per minute and as the number of bursts per 100 heart beats, to correct for differences in heart rate.
Resting sympathetic activity | Post partum (6-10 weeks after delivery)
  Resting sympathetic activity is measured by microneurography, as expressed as the number of bursts per minute and as the number of bursts per 100 heart beats, to correct for differences in heart rate.
Serum corin content measurement | Early pregnancy (< 12 weeks gestation)
  Serum corin content will be measured by venous blood samples
Serum corin content measurement | Late pregnancy (30-34 weeks of gestation)
  Serum corin content will be measured by venous blood samples
Serum corin content measurement | Post partum (6-10 weeks after delivery)
  Serum corin content will be measured by venous blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Qi Fu, MD, PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (2):
- United States (2):
  - Institute for Exercise and Environment Medicine (IEEM) at Texas Health Presbyterian Hospital, Dallas, Texas
  - University of Texas Southwestern Medical Center Dallas, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No